CLINICAL TRIAL: NCT00473369
Title: Prognosis of Atypical Pituitary Adenomas
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tohoku University (Other)
Other Study IDs: 1-2007.nsg.med.tohoku
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2007-05

CONDITIONS: Pituitary Diseases
Keywords: atypical adenoma; Ki-67; p53; pituitary; prognosis
MeSH Terms: conditions — Pituitary Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Context: Pituitary adenoma is generally indolent, but an aggressive subtype called atypical adenoma has uncertain prognosis, and an unclear relationship between prognosis and morphology.

Objective: This study investigated the prognostic factors of this tumor. Design: Retrospective analysis. Setting: University and associated hospitals.

ELIGIBILITY:
Inclusion Criteria:

* pituitary adenomas of more than 3 % of Ki67 labeling index surgically treated at Tohoku university and associated hospital

Exclusion Criteria:

* pituitary adenomas of less than 3 % of Ki-67 labeling index surgically treated at Tohoku university and associated hospital

Ages: 12 Years to 74 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-01; Study Completion 2007-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshikazu Ogawa, M. D., Principal Investigator — Department of neurosurgery, Tohoku university